CLINICAL TRIAL: NCT01394185
Title: Effects of Dronabinol (Oral THC) on Cannabis Use
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00041251; R01DA025044 (NIH)
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Marijuana Smoking
Keywords: marijuana; dronabinol; pharmacotherapy
MeSH Terms: conditions — Marijuana Smoking; Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Dose Dronabinol, High Dose Dronabinol, and placebo (Active Comparator): Participants were administered dronabinol (0 mg/day, 120mg/day and 240mg/day) for 12 days each in a random order
  Interventions: Drug: Dronabinol 120mg/day; Drug: Placebo; Drug: Dronabinol 240mg/day

INTERVENTIONS:
Drug: Dronabinol 120mg/day — Participants receive 40mg dronabinol 3 times daily
  Other Names: Marinol; THC
Drug: Placebo — Participants receive placebo
Drug: Dronabinol 240mg/day — Participants receive 80mg dronabinol 3 times daily
  Other Names: Marinol; THC

SUMMARY:
Study participants received dronabinol (0, 120mg/day and 240mg/day) for 12 consecutive days in a randomized order. During each dronabinol maintenance period they were able to self-administer active or placebo cannabis using either a progressive ratio schedule or choice between cannabis and monetary alternative.

ELIGIBILITY:
Inclusion Criteria:

* Current use of marijuana
* Able to give informed consent

Exclusion Criteria:

* Daily use of psychoactive medication
* Current Axis I psychiatric disorder other than dependence on cannabis or nicotine, or abuse of drugs or alcohol
* Women who are pregnant, breast feeding, or planning to become pregnant within the next 3 months
* Those seeking treatment for cannabis-related problems or using cannabis under the guidance of a physician for a medical disorder
* Uncontrolled or unstable cardiovascular disease
* Allergy to sesame oil

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (Bayview Campus), Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, 120mg, 240mg; 120mg, 240mg, Placebo; 240mg, 120mg, Placebo; 120mg, Placebo, 240mg; 240mg, Placebo, 120mg; Placebo, 240mg, 120mg: Participants received dronabinol for 12 days in the above order in a within-subject crossover
Period: Overall Study
Arm/Group | Placebo, 120mg, 240mg | 120mg, 240mg, Placebo | 240mg, 120mg, Placebo | 120mg, Placebo, 240mg | 240mg, Placebo, 120mg | Placebo, 240mg, 120mg
Started | 8 | 2 | 2 | 4 | 6 | 3
Completed | 2 | 2 | 2 | 3 | 2 | 2
Not Completed | 6 | 0 | 0 | 1 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Change in protocol | 3 | 0 | 0 | 0 | 3 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants received dronabinol (PL, 120mg, 240mg/day) in a randomized within-subject crossover design
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Marijuana Self-administration - Progressive Ratio
Description: Participants will be able to self-administer cannabis cigarettes (weighing about 0.8 grams and with about 6% THC) under a progressive ratio schedule. The number of progressive ratios completed (and thus, cannabis cigarettes consumed) is the primary study endpoint
Time Frame: 12-day Dronabinol maintenance period
Measure: Mean (Standard Error); unit: Progressive Ratios Completed
Groups:
- Placebo: Placebo maintenance period
- 120mg Dronabinol: 120mg/day (40mg tid) dronabinol maintenance period
- 240mg Dronabinol: 240mg/day (80mg tid) dronabinol maintenance period
Arm/Group | Placebo | 120mg Dronabinol | 240mg Dronabinol
Number analyzed (Participants) | 13 | 13 | 13
Progressive Ratios Completed | 5.2 (0.2) | 4.5 (0.2) | 4.4 (0.2)

2. Primary Outcome: Marijuana Self-administration - Drug Vs Money Choice
Description: Participants will be able to self-administer cannabis cigarettes (weighing about 0.8 grams and with about 6% THC) in 5 discrete choices each day between one cannabis cigarette and $1. The number of cannabis cigarettes chosen (and subsequently self-administered) is the primary study endpoint
Time Frame: 12-day Dronabinol maintenance period
Measure: Mean (Standard Error); unit: Cannabis Cigarettes Chosen
Arm/Group | Placebo | 120mg Dronabinol | 240mg Dronabinol
Number analyzed (Participants) | 13 | 13 | 13
Cannabis Cigarettes Chosen | 3.5 (0.6) | 2.3 (0.4) | 2.5 (0.5)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Placebo: Placebo dronabinol maintenance
- 120mg Dronabinol: 120mg (40mg tid) dronabinol maintenance
- 240mg Dronabinol: 240mg (80mg tid) dronabinol maintenance
Arm/Group | Placebo | 120mg Dronabinol | 240mg Dronabinol
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes